CLINICAL TRIAL: NCT04778254
Title: PEEK Versus Metallic Attachment-retained Obturators Regarding Patient Satisfaction: A Randomized Controlled Trial.
Brief Title: PEEK Versus Metallic Attachment-retained Obturators
Acronym: PEEK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sharaf Mohamed Yahia, Principal Investigator,, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 38/10/2018
Record Dates: First submitted 2021-02-22; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Maxillary Neoplasms
MeSH Terms: conditions — Maxillary Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- conventional obturator (Active Comparator): conventional group received conventional clasp-retained obturators with metallic framework (Control group).
  Interventions: Other: conventional obturator
- metallic attachment retained obturator (Experimental): metal group received an attachment-retained obturator with metallic framework
  Interventions: Other: metalic attachment retained obturator
- PEEk attachment retained obturator (Experimental): PEEK group received attachment-retained obturators with milled PEEK framework,
  Interventions: Other: PEEK attachment retained obturator

INTERVENTIONS:
Other: PEEK attachment retained obturator — attachment retained obturator for management of hemi maxillectomy
  Other Names: milled PEEK obturator
  Arms: PEEk attachment retained obturator
Other: metalic attachment retained obturator — attachment retained obturator for management of hemi maxillectomy
  Other Names: attachment retained obturator
  Arms: metallic attachment retained obturator
Other: conventional obturator — clasp retained obturator for management of hemi maxillectomy
  Other Names: clasp retained obturator
  Arms: conventional obturator

SUMMARY:
Patients' satisfaction evaluation and radiographic evaluation of the terminal abutments of attachment- retained maxillary obturators with metal framework versus milled PEEK framework in the management of maxillectomy cases.

DETAILED DESCRIPTION:
Eighteen participants were randomly divided into three parallel groups (n=6). Participants of PEEK group received attachment-retained obturators with milled PEEK framework, metal group received an attachment-retained obturator with metallic framework and conventional group received conventional clasp-retained obturators with metallic framework (Control group). Evaluation included radiographic evaluation and patients' satisfaction where two scales were followed in this study, including "The Obturator Functioning Scale" and "The European Organization for Research and Treatment of Cancer Head and Neck 35" using one way ANOVA test.

ELIGIBILITY:
Inclusion Criteria:

* patient underwent surgical removal of half of maxilla
* participants with a sufficient number of natural teeth(class I and \or class IV Aramany classification) not less than 5 teeth, mouth opening is not less than 25 mm, intact soft palate,

Exclusion Criteria:

* participants are exposed to radiotherapy or chemotherapy during last year.
* participant with congenital defect

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
patient satisfaction 1(change" is being assessed) | 1 week to 6 months
  The Obturator Functioning Scale ( minimum value is "1"and maximum value is "5"
patient satisfaction 2 (change" is being assessed) | 1 week to 6 months
  The European Organization for Research and Treatment of Cancer Head and Neck 35 ( minimum value is "1"and maximum value is "5"

SECONDARY OUTCOMES:
Radiographic evaluation (change" is being assessed) | base line,6 months, 9 months,12 months
  evaluation of terminal abutment

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Sharaf, lecturer, Principal Investigator — Beni-Suef University
Locations (1):
- Mohamed Sharaf, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
finished work will be published